CLINICAL TRIAL: NCT02035111
Title: To Evaluate the Safety and the Efficacy of Tianshu Capsule Treating Migraine in a Randomized, Placebo-Controlled, Double-blind, Multicenter Study.
Brief Title: A Randomized, Placebo-Controlled, Double-blind Study of Tianshu Capsule in the Treatment of Migraine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Bionovo Medicine Development Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z-TSJN-JN-Ⅳ
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Migraine
Keywords: Migraine; Tianshu capsule
MeSH Terms: conditions — Migraine Disorders | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tianshu capsule (Experimental): Four Tianshu capsules (0.34 g per capsule) by oral three times a day for 12 weeks.
  Interventions: Drug: Tianshu capsule
- Sugar pill (Placebo Comparator): Four sugar pills (0.34 g per capsule) by oral three times a day for 12 weeks.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Tianshu capsule
  Arms: Tianshu capsule
Drug: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of Tianshu capsule treating Migraine Headache.

DETAILED DESCRIPTION:
Primary headache disorders,particularly migraine is globally prevalent. Many studies show the burdens they impose: pain, disability, reduced quality of life (QoL), marked impairment of participation in work and social activities, and heavy financial costs.

The purpose of this study is to evaluate the safety and the efficacy of Tianshu capsule treating Migraine Headache. To provide a safe and effective treatment of Migraine Headache.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the Migraine diagnosis.
* Age of onset should be before age 50 years.
* Migraine must have been occurring for 1 year preceding entry into the trial.
* The number of migraine attack should be no less than 6 for a period of 3 months prior to Screening stage.
* The number of migraine days is to be 2-8 for a period of 1 month prior to screening for entry into the trial.
* Migraine days should be less than 15 for a period of 1 month prior to screening for entry into the trial.
* Ages 18-65.
* Participant can understand and complete the Headache diary.
* All participants signed the informed consent.

Exclusion Criteria:

* Other migraine prophylactic medication is continued 3 months prior to the drug trial.
* Participants who have taken Tianshu capsule during 1 month prior to Screening stage.
* The number of acute treatment for migraine is more than 10 per month.
* Participants who have taken antipsychotics or antidepressant medications (unless only for migraine prophylaxis) during the previous 3 months.
* Participants who abuse alcohol or other drugs.
* Participants who are resistant to all acute migraine drugs prescribed optimally.
* hypotension or uncontrolled hypertension.
* Severe infections.
* Malignancy.
* Significant medical history of such as cardiac disease, cerebrovascular disease, liver disease, nephropathy etc.
* Known allergies or serious side effects with Tianshu capsule in the past.
* Breastfeeding, pregnant and potentially fertile women participant.
* History of cluster headaches, tension-type headache, vascular headache with non-migraine, drug - dependence headache.
* Secondary headaches, including hypertension, post-traumatic brain syndrome etc.
* Participants who have taken migraine prophylactic medication regularly during 1 month prior to Screening stage.
* Participants who are taking part in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 947 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of attack of Migraine Per 4 weeks at Week 16 from baseline | -4w,0,4w,8w,12w,16w

SECONDARY OUTCOMES:
Change in seizure duration of Migraine Per 4 weeks at Week 16 from baseline. | -4w,0,4w,8w,12w,16w
Change in degree of pain of Migraine Per 4 weeks at Week 16 from baseline. | -4w,0,4w,8w,12w,16w
Change in the days using acute therapy of Migraine Per 4 weeks at Week 16 from baseline. | -4w,0,4w,8w,12w,16w
Proportion of subjects whose number or days of migraine attacks reduce at least 50%. | -4w,0,4w,8w,12w,16w
Change in number of concomitant migrainous symptoms attacks Per 4 weeks at Week 16 from baseline. | -4w,0,4w,8w,12w,16w
Safety assessments will be based on adverse event reports and the results of vital sign measurements, electrocardiogram, and clinical laboratory tests. | 0, 12w
  Adverse event reports will be assessed at 0, 4w, 8w, 12w, 16w. clinical laboratory tests including WBC, RBC, HGB, PLT, LEU, ERY, PRO,Stool routine, ALT, AST, TBil, ALP, GGT, BUN, Cr will be assessed at 0, 12w.
  Electrocardiogram will be assessed at 0, 12w. Vital sign measurements will be assessed at -4w, 0, 4w, 8w, 12w, 16w.

CONTACTS AND LOCATIONS:
Overall Officials: Shengyuan Yu, Principal Investigator — Chinese PLA General Hospital
Locations (20):
- China (20):
  - The People's Hospital,Huaibei, Huaibei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Daxing hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Quanzhou First Hospita, Quanzhou, Fujian
  - SanMing First Hospital, Sanming, Fujian
  - The People's Hospital,Cangzhou, Cangzhou, Hebei
  - Langfang hospital of Traditional Chinese Medicine, Langfang, Hebei
  - The two six zero hospital of Chinese people's Liberation Army, Shijiazhuang, Hebei
  - Tangshan TCM Hospital, Tangshan, Hebei
  - Kaifeng hospital of Traditional Chinese Medicine, Kaifeng, Henan
  - Luohe hospital of Traditional Chinese Medicine, Luohe, Henan
  - Wuhan sixth hospital, Wuhan, Hubei
  - Yiyang central hospital, Yiyang, Hunan
  - The Affiliated Hospital of Changchun University of Chinese medicine, Changchun, Jilin
  - Jilin brain hospital, Siping, Jilin
  - Jinan hospital of traditional Chinese Medicine, Jinan, Shandong
  - The second affiliated hospital of Shandong Traditional Chinese Medicine University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Jining First Hospital, Jining, Shandong
  - Xi An Hospital of Traditional Chinese Medicine, Xian, Shanxi

REFERENCES:
- [Derived] Yu S, Ran Y, Xiao W, Tang W, Zhao J, Chen W, Zhuang H, Ouyang C, Lin H, Liu D, Chen T, Huang H, Wang B, Hao Y, Yan Z, Zhao S, Wang Y, Ni J, Wang C, Ding W, Li G, Cao J, Tian S. Treatment of migraines with Tianshu capsule: a multi-center, double-blind, randomized, placebo-controlled clinical trial. BMC Complement Altern Med. 2019 Dec 16;19(1):370. doi: 10.1186/s12906-019-2775-2. PMID 31842860